CLINICAL TRIAL: NCT06978569
Title: A Randomized, Outcome Assessor-Blinded Clinical Trial Comparing the Efficacy of Acellular Dermal Matrix (ADM) Hydrogel Versus Alginate Dressings in the Treatment of Chronic Traumatic Wounds
Brief Title: Comparative Efficacy of ADM Hydrogel vs. Alginate Dressings in Chronic Trauma Wounds
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fateme Abedini, Principal Investigator, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IR.ARI.MUI.REC.1404.054
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Trauma Wounds
Keywords: chronic wound; acellular dermal matrix; ADM; wound size; alginate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In addition to outcome assessors, the data analyst is blinded to the randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADM hudrogel group (Experimental): Participants in this group will receive an acellular dermal matrix (ADM) hydrogel applied directly to the wound bed following standard debridement procedures. After application, the wound will be covered with a standard secondary dressing. Dressing changes will be performed every 2 to 3 days, or as clinically indicated based on wound condition and healing progress.
  Interventions: Device: Injectable Acellular dermal matrix hydrogel
- Alginate Dressing Group (Active Comparator): Participants in this group will receive an alginate dressing applied directly to the wound bed following debridement. The wound will be managed with dressing changes performed according to the manufacturer's instructions and standard clinical protocol.
  Interventions: Device: Alginate dressing

INTERVENTIONS:
Device: Injectable Acellular dermal matrix hydrogel — An injectable, sterile acellular dermal matrix (ADM) gel derived from processed biological tissue, designed to promote healing in chronic wounds. The gel is injected directly onto the wound bed following standard debridement and serves as a biocompatible scaffold to support granulation tissue formation, epithelialization, and wound closure. After application, the wound is covered with a standard secondary dressing. Dressing changes are performed every 2 to 3 days or as clinically indicated.
  Arms: ADM hudrogel group
Device: Alginate dressing — A sterile, absorbent alginate wound dressing composed of natural polysaccharide fibers derived from seaweed. Following standard debridement, the alginate dressing is applied directly to the wound bed to manage exudate and maintain a moist wound environment conducive to healing. The dressing is covered with a secondary dressing and changed according to the manufacturer's instructions and clinical protocol.
  Arms: Alginate Dressing Group

SUMMARY:
The goal of this clinical trial is to find out whether a wound treatment made from acellular dermal matrix (ADM) gel can help heal chronic traumatic wounds more effectively than standard alginate dressings in adults aged 18 and older with wounds that have lasted more than 3 weeks.

The main questions it aims to answer are:

Does ADM gel reduce the size of chronic wounds more than alginate dressings after 12 weeks?

Does ADM gel help wounds heal faster and improve quality of life for patients?

Researchers will compare ADM gel to alginate dressings to see if the ADM gel leads to better healing results and fewer complications.

Participants will:

Be randomly assigned to receive either ADM gel or alginate dressing.

Have the treatment applied directly to their cleaned wound.

Attend weekly visits for up to 12 weeks for wound checks, measurements, and dressing changes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic trauma wounds persisting ≥3 weeks.
* Wound size between 4 and 20 cm² and depth ≤9 mm on the lower limbs.
* Willingness and ability to provide informed consent.
* Wounds without uncontrolled infection

Exclusion Criteria:

* Wounds with exposed bone.
* Current use of immunomodulators, corticosteroids, immunosuppressive or cytotoxic drugs.
* Pregnant individuals.
* Significant reduction (≥30%) of wound size during a 2-week run-in phase.
* Concurrent participation in another clinical trial involving drugs.
* Wounds with uncontrolled infection
* Allergy or hypersensitivity to components of ADM gel or alginate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Wound surface area (cm²) at Week 12, adjusted for baseline wound size | Week 1 and 12
  Wound surface area is measured as length × width (in cm²) using digital planimetry. Comparison of wound size between groups at Week 12 will be conducted using ANCOVA, adjusting for baseline wound size and relevant covariates.

SECONDARY OUTCOMES:
Time to complete wound healing (100% epithelialization) | Weekly up to 12 weeks
  Number of days from baseline to full wound closure, defined as 100% epithelialization with no drainage.
Rate of granulation tissue formation | Weekly up to 12 weeks
  Visual and digital assessment of granulation tissue coverage over time.
Rate of wound epithelialization | Weekly up to 12 weeks
  Proportion of wound area covered by new epithelium, assessed at each follow-up visit.
Incidence of complications (infection, necrosis, bleeding) | Up to 12 weeks
  Number and type of wound-related adverse events recorded during follow-up.
Quality of life score at Week 12 | Weeks 1 and 12
  Patient-reported quality of life is assessed using the SF-36 questionnaire at baseline and Week 12. Group differences at Week 12 will be analyzed using ANCOVA, adjusting for baseline SF-36 scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Alzahra hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR, Analytic Code
Access Criteria: Individual participant data (IPD) underlying published results will be available upon reasonable request from qualified researchers with a methodologically sound proposal.